CLINICAL TRIAL: NCT07391306
Title: Double-blind, Placebo-controlled, Adaptive, Multicenter, Prospective, Randomized, Comparative, Parallel-group Study of the Efficacy and Safety of Neovasculgen (Plasmid Supercoiled Deoxyribonucleic Acid pCMV-VEGF165) in Painful Bladder Syndrome/Interstitial Cystitis (BPS/IC)
Brief Title: The Study is Being Conducted to Find a New Treatment for Patients Suffering From Interstitial Cystitis Without Hunner's Lesions.
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: JSC NextGen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-InterCis-NVG-III
Record Dates: First submitted 2026-01-13; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: IC; Interstitial Cystitis and Bladder Pain Syndrome; Interstitial Cystitis, Chronic
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The investigational therapy group (Experimental): Receiving combination therapy: coagulation of Hunner's lesions of the bladder followed by hydrobougienage and intradetrusor administration of Neovasculgen
  Interventions: Drug: Neovasculgen®
- Placebo group (Placebo Comparator): Control group, receiving basic therapy: coagulation of Hunner's lesions of the bladder followed by hydrobougienage
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neovasculgen® — The bladder is hydro-bougienaged, followed by intradetrusor injections using a cystoscopic injection needle inserted into a rigid or flexible cystoscope inserted through the urethra into the bladder, under direct visualization. The drug is administered as 30 injections, evenly throughout the bladder.
  Arms: The investigational therapy group
Drug: Placebo — The bladder is hydro-bougienaged, followed by intradetrusor injections using a cystoscopic injection needle inserted into a rigid or flexible cystoscope inserted through the urethra into the bladder, under direct visualization. The drug is administered as 30 injections, evenly throughout the bladder.
  Arms: Placebo group

SUMMARY:
To evaluate the efficacy and safety of Neovasculgen in interstitial cystitis and the prevention of secondary bladder shrinkage with a decrease in its volume.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to any study-related procedures.
2. Women aged 18 to 65 years, inclusive.
3. A confirmed diagnosis of painful bladder syndrome/interstitial cystitis, characterized by pelvic pain associated with filling or emptying the bladder, frequent urination day and night, with symptoms lasting at least 12 months, with the exclusion of a urinary tract infection or other disease that could cause such symptoms.
4. Absence of Hunner's lesions of the bladder during cystoscopy with hydrobougienage of the bladder (2 minutes, 80 cm H2O).
5. A glycated hemoglobin level within the normal range for the patient's age group.
6. Ability to comply with all study requirements, at the discretion of the investigator, including regularly keeping a voiding diary, completing questionnaires, and attending all scheduled study visits.
7. Women who are of childbearing potential must have negative pregnancy test results and must use reliable contraception throughout their participation in the study.

Exclusion Criteria:

1. Any condition that prevents intravesical administration of medications.
2. Received medication or non-medication therapy, including physical therapy, for BPS/IC within 1 month prior to study inclusion.
3. Instillation of any pharmacological agent into the bladder less than 1 month prior to screening.
4. History of chronic drug or alcohol abuse.
5. Pregnant women, planning to become pregnant during the study, or currently breastfeeding.
6. Any other conditions associated with pelvic pain, except for BPS
7. Pelvic surgery less than 6 months prior to the study
8. Any intravesical procedures, except for diagnostic cystoscopy, less than 3 months prior to screening
9. History of allergy or intolerance to the anesthetic or antibiotics that the investigator intends to use during the study.
10. Inability to discontinue anticoagulant/antiplatelet medications at least 5 days prior to each investigational drug administration and resume them on the 4th day after each investigational drug administration (low molecular weight heparin may be used for 3 days after investigational drug administration).
11. Diseases of the urinary tract/bladder (neoplasms, tuberculous and bacterial cystitis, urolithiasis, radiation injury, urethral diverticulum, neurogenic dysfunction of the lower urinary tract) and female genital organs (neoplasms, vaginitis, genital infections).
12. Other conditions that, in the opinion of the research physician, could become an objective obstacle to the patient's participation in the study and/or create additional risks for the patient.
13. A history of intravesical botulinum therapy performed within the last 12 months prior to inclusion in this study.
14. Bladder capacity under anesthesia less than 150 ml.
15. Residual urine volume greater than 50 ml.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
"Number of Participants with Treatment-Related effect according to the protocol through study completion, on average, over 1 year. | Until the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Botkin Hospital, Moscow, Russia